CLINICAL TRIAL: NCT00316745
Title: Irinotecan Combined With S-1( IRIS ) Followed by mFOLFOX6 Regimen Versus mFOLFOX6 Followed by IRIS Regimen in Advanced Colorectal Cancer
Brief Title: IRIS Followed by mFOLFOX6 or the Reverse Sequence in Advanced Colorectal Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Because of approval of Bevacizumab, it was difficult to perform clinical study in 1st line setting.
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0601; IFOX study
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: irinotecan; S-1; Oxaliplatin; l-leucovorin; Fluorouracil; Metastatic colorectal cancer; phase III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; titanium silicide; S 1 (combination); Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): mFOLFOX6 （ → IRIS ( Irinotecan and S-1) ）
  Interventions: Drug: L-Plat; Drug: Isovorin; Drug: 5-FU
- 2 (Experimental): IRIS ( Irinotecan and S-1 ) → mFOLFOX6
  Interventions: Drug: Campto, Topotesin; Drug: TS-1

INTERVENTIONS:
Drug: Campto, Topotesin — 100 mg/m2, IV (in the vein) on day 1,15 of each cycle.
  Other Names: Irinotecan
  Arms: 2
Drug: TS-1 — S-1 Day1~14, everyday P.O.(Day 15~28 rest)
  Other Names: S-1
  Arms: 2
Drug: L-Plat — Oxaliplatin (85mg/m2) Day 1, 15
  Other Names: Oxaliplatin
  Arms: 1
Drug: Isovorin — l-leucovorin (200mg/m2) Day 1, 15
  Other Names: l-leucovorin
  Arms: 1
Drug: 5-FU — 400 mg/m2, IV (in the vein) on day 1,15 of each 28 day cycle. 2400 mg/m2, CIV (in the vein) on day 1~3 (48 hours) of each 28 day cycle.
  Other Names: Fluorouracil
  Arms: 1

SUMMARY:
This randomized phase III study compares safety and efficacy of two sequence arms in advanced colorectal cancer: irinotecan and S-1 (IRIS) followed by oxaliplatin containing regimen (arm A), or l-leucovorin (l-LV), 5-FU and oxaliplatin (mFOLFOX6) followed by irinotecan containing regimen (arm B).

DETAILED DESCRIPTION:
A multicenter randomized open-label controlled phase III study is conducted in patients with inoperable advanced or metastatic colorectal cancer who receive no previous chemotherapy. Usefulness of IRIS and mFOLFOX6 regimens as the 1st-line therapy for colorectal cancer is evaluated in PFS, MST, incidence and severity of adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of colorectal cancer. 2） Age: 18 - 75 years. 3） No prior chemotherapy 4） ECOG Performance Status 0 to 2 5) A life expectancy of at least 3 months 6) Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC ≧3,500/mm3 and Neutrophil ≧2,000/mm3. Hb ≧10.0 g/dl. Platelet count ≧100,000/mm3. AST and ALT ≦2.5 times the upper limit of normal (excluding liver metastasis). T-Bil ≦1.5 mg/dl. Creatinine ≦1.5 mg/ dl. 7).Patients must have the ability to understand and the willingness to sign a written informed contact document.

Exclusion Criteria:

1. Patients receiving blood transfusion, blood derivatives or granulocyte-colony stimulating factor within 7days prior to entering the study.
2. Patients can not have oral intake
3. Patients receiving Flucytosine treatment
4. Patients with severe pleural effusion or ascites.
5. Patients who have brown brain metastasis
6. Patients with diarrhea 4 or more times per day
7. Patients with active gastrointestinal bleeding.
8. Patients with intestinal obstruction
9. Patients with active infection.
10. Patients with serious pulmonary disease (such as interstitial pneumonia, pulmonary fibrosis, pulmonary emphysema)
11. Patients with serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
12. Patients with significant cardiac disease.
13. Patients with active multiple cancer.
14. Patients with neuropathy ≥ grade 2
15. Patients who are pregnant, are of childbearing potential, or breast-feeding.
16. Patients with severe mental disorder.
17. Patients with a history of serious allergic reaction.
18. Judged to be ineligible for this protocol by the investigation.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-04; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
PFS of 1st line treatment | 2-years

SECONDARY OUTCOMES:
OS | 4-years
objective tumor response | 1-year
PFS of 2nd line treatment | 1-year
safety | 4-years

CONTACTS AND LOCATIONS:
Overall Officials: Yoshito Komatsu, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital (Hokkaido University Graduate School of Medicine / School of Medicine), Sapporo, Hokkaido, Japan